CLINICAL TRIAL: NCT03804879
Title: A Randomized Patient-and-physician Blinded, Placebo-controlled, 24-week Study to Assess the Safety, Tolerability and Efficacy of LMB763 in Patients With Diabetic Nephropathy
Brief Title: Safety, Tolerability and Efficacy of Nidufexor in Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLMB763X2202; 2018-002491-40 (EudraCT Number)
Record Dates: First submitted 2018-11-26; First posted 2019-01-15 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Nephropathy
Keywords: diabetes
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LMB763 (Experimental): 50 mg LMB763 (two LMB763 25 mg capsules) were orally administered once daily for 24 weeks in addition to SoC.
  Interventions: Drug: Nidufexor; Drug: Standard of Care (SoC)
- Placebo (Placebo Comparator): Placebo was orally administered once daily for 24 weeks in addition to SoC.
  Interventions: Other: Placebo; Drug: Standard of Care (SoC)

INTERVENTIONS:
Drug: Nidufexor — 50 mg (two 25 mg) LMB763 capsules for oral administration
  Other Names: LMB763
  Arms: LMB763
Other: Placebo — Placebo capsules for oral administration
  Arms: Placebo
Drug: Standard of Care (SoC) — Optimal tolerated doses of angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB)

SUMMARY:
Nidufexor addresses fibrosis, oxidative stress, inflammation and cell death, and therefore has the potential to improve the management of diabetic kidney disease when added to the standard of care (SoC) (angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB)).

This non-confirmatory Phase 2 study was designed to determine the safety, tolerability, efficacy, pharmacokinetics and pharmacodynamics of nidufexor in combination with ACEI or ARB at a dose level that is SoC as judged by the study doctor in patients with type 2 diabetes and nephropathy.

DETAILED DESCRIPTION:
This was a non-confirmatory, multicenter, patient- and investigator-blinded, randomized, and placebo-controlled, proof-of concept trial assessing nidufexor vs. placebo in patients receiving standard of care (optimal tolerated doses of ARB or ACEI) for diabetic nephropathy due to type 2 diabetes.

The study consisted of three distinct study periods:

Screening (Day -30 to Day-1): lasted up to a maximum of 30 days and comprised a screening / baseline assessment. This visit was used to confirm that the study inclusion and exclusion criteria were met and served as baseline assessment prior to randomization. Participant randomization occurred prior to day 1 as soon as participant eligibility was confirmed.

Treatment period (Day 1-168): Participants were randomized in a 1:1 ratio to receive nidufexor 50 mg or placebo once daily for 24 weeks. Nidufexor and placebo were given in addition to SoC (optimal tolerated doses of ARB or ACEI).

End of Study (EOS) and Safety follow-up (Day 169 to Day 197): Study assessments were performed until the EOS visit (Day 169). Post Study Safety Contact occurred approximately 28 days after discontinuing study treatment until day 197.

ELIGIBILITY:
Inclusion Criteria:

* Male/female patients, 18-75 years
* Written informed consent
* Diagnosis of Type 2 diabetes mellitus, with diagnosis made at least 6 months prior to screening
* Diabetic nephropathy as evidenced by Urine albumin-Cr ratio (UACR) ≥300 mg/g Cr at screening while receiving a dose of angiotensin converting enzyme inhibitor or angiotensin receptor blocker that is the standard of care as judged by the study doctor.

Exclusion Criteria:

* History of type 1 diabetes mellitus
* Severe renal impairment manifesting as serum creatinine eGFR < 30 mL/min/1.73 m^2 at screening
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, unless they are using basic methods of contraception during dosing of study treatment
* Uncontrolled diabetes mellitus at screening
* History or current diagnosis of ECG abnormalities prior to first study dose
* History of kidney disease other than diabetic nephropathy at screening
* Uncontrolled hypertension at screening
* Use of prohibited medications, including but not limited to GLP-1 agonists and SGLT2 inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (5):
  - Novartis Investigative Site, Miami Lakes, Florida
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Norman, Oklahoma
  - Novartis Investigative Site, El Paso, Texas
  - Novartis Investigative Site, Sugar Land, Texas
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Novartis Investigative Site, Prague, Czechia
- Germany (3):
  - Novartis Investigative Site, Essen, Nordrhine Westphalia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Elsterwerda
- Novartis Investigative Site, Amman, Jordan
- Lebanon (2):
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Saida
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Talas / Kayseri

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 18 sites in 7 countries.
Pre-assignment Details: Participants underwent a Screening period of up to 30 days which included screening and baseline assessments.
Period: Overall Study
Arm/Group | LMB763 | Placebo
Started (All randomized participants.) | 41 | 42
Pharmacokinetics (PK) Analysis Set (All randomized participants with at least one valid PK concentration measurement, who received LMB763 and no protocol deviations with relevant impact on PK data.) | 41 | 0
Pharmacodynamics (PD) Analysis Set (All randomized participants with no protocol deviations with relevant impact on PD data.) | 41 | 41
Completed | 25 | 29
Not Completed | 16 | 13
Not completed — Adverse Event | 3 | 0
Not completed — Study Terminated By Sponsor | 10 | 12
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LMB763 | Placebo | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (8.95) | 61.6 (8.36) | 61.2 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 28 | 32 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 41 | 41 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ratio to Baseline in Urinary Albumin to Creatinine Ratio (UACR)
Description: UACR is a ratio between albumin and creatinine, and it estimates 24-hour urine albumin excretion.
  UACR (mg/mmol) = urine albumin [mg/L] / urine creatinine [mmol/L]. UACR was analyzed on a log-scale fitting a repeated measures mixed model including treatment and visit as fixed effects and log of baseline as continuous covariate. Baseline is the last measurement prior to treatment administration. No methods for imputation of missing data were used. Values reported were back-transformed to original scale. A lower score in the ratio to baseline indicates improvement.
Time Frame: Baseline and days 14, 29, 57, 85, 113, 141 and 169
Population: All randomized participants. At each time point, only participants with a value at both baseline and that time point were included.
Measure: Least Squares Mean (80% Confidence Interval); unit: Ratio to baseline
Arm/Group | LMB763 | Placebo
Number analyzed (Participants) | 41 | 42
Ratio to baseline
  Day 14: number analyzed (Participants) | 39 | 42
  Day 14 | 0.90 [0.79 to 1.02] | 1.06 [0.94 to 1.20]
  Day 29: number analyzed (Participants) | 37 | 39
  Day 29 | 0.83 [0.75 to 0.93] | 1.00 [0.90 to 1.12]
  Day 57: number analyzed (Participants) | 34 | 35
  Day 57 | 0.85 [0.76 to 0.94] | 1.05 [0.95 to 1.17]
  Day 85: number analyzed (Participants) | 29 | 35
  Day 85 | 0.84 [0.72 to 0.97] | 1.07 [0.93 to 1.23]
  Day 113: number analyzed (Participants) | 26 | 30
  Day 113 | 0.87 [0.73 to 1.04] | 1.07 [0.90 to 1.26]
  Day 141: number analyzed (Participants) | 23 | 27
  Day 141 | 0.84 [0.71 to 1.01] | 1.15 [0.98 to 1.35]
  Day 169: number analyzed (Participants) | 26 | 30
  Day 169 | 0.74 [0.61 to 0.89] | 0.92 [0.78 to 1.10]

2. Primary Outcome: Ratio to Baseline in 24 Hour Urinary Albumin at Week 24 (Day 169)
Description: Albuminuria describes the existence of albumin in the urine and the gold-standard to assess albuminuria is 24-hour urinary albumin excretion (milligram/24 hours). An analysis of covariance (ANCOVA) with treatment as the classification factor and log-transformed baseline as the covariate was conducted for log-transformed ratio to baseline 24-hour urinary albumin excretion. Baseline is the last measurement prior to treatment administration. No methods for imputation of missing data were used. Values reported were back-transformed to original scale. A lower score in the ratio to baseline indicates improvement.
Time Frame: Baseline and day 169
Population: Pharmacodynamics (PD) analysis set. Only participants with a value at both baseline and at Day 169 were included.
Measure: Least Squares Mean (80% Confidence Interval); unit: Ratio to baseline
Arm/Group | LMB763 | Placebo
Number analyzed (Participants) | 17 | 21
Ratio to baseline | 0.58 [0.45 to 0.74] | 0.91 [0.72 to 1.14]

3. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with AEs and SAEs including significant changes from baseline in vital signs, electrocardiograms and laboratory values qualifying and reported as AEs. The category Number of participants with AEs includes also the number of participants with SAEs. The number of participants in each category is reported in the table.
Time Frame: From the start of treatment to 28 days after end of treatment, assessed up to maximum duration of 197 days
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | LMB763 | Placebo
Number analyzed (Participants) | 41 | 42
Participants
  AEs | 29 | 25
  SAEs | 2 | 2

4. Secondary Outcome: Ratio to Baseline in Estimated Glomerular Filtration Rate (eGFR)
Description: Estimate Glomerular Filtration Rate (GFR) calculates estimated GFR (eGFR) from serum creatinine levels to assess kidney function. eGFR (milliliter/minute) was analyzed on a log-scale fitting a repeated measures mixed model including treatment and visit as fixed effects and log of baseline as continuous covariate. Baseline is the last measurement prior to treatment administration. No methods for imputation of missing data were used. Values reported were back-transformed to original scale. A higher score in the ratio to baseline indicates improvement.
Time Frame: Baseline and days 14, 29, 57, 85, 113, 141 and 169
Population: Pharmacodynamics (PD) analysis set. At each time point, only participants with a value at both baseline and that time point were included.
Measure: Least Squares Mean (80% Confidence Interval); unit: Ratio
Arm/Group | LMB763 | Placebo
Number analyzed (Participants) | 41 | 41
Ratio
  Day 14: number analyzed (Participants) | 38 | 41
  Day 14 | 0.95 [0.93 to 0.98] | 0.96 [0.94 to 0.99]
  Day 29: number analyzed (Participants) | 36 | 37
  Day 29 | 0.94 [0.91 to 0.97] | 0.94 [0.91 to 0.97]
  Day 57: number analyzed (Participants) | 32 | 32
  Day 57 | 0.98 [0.95 to 1.02] | 0.96 [0.93 to 1.00]
  Day 85: number analyzed (Participants) | 28 | 32
  Day 85 | 0.97 [0.93 to 1.01] | 0.94 [0.90 to 0.97]
  Day 113: number analyzed (Participants) | 26 | 23
  Day 113 | 0.96 [0.92 to 0.99] | 0.94 [0.91 to 0.98]
  Day 141: number analyzed (Participants) | 22 | 23
  Day 141 | 0.98 [0.95 to 1.02] | 0.93 [0.90 to 0.96]
  Day 169: number analyzed (Participants) | 21 | 25
  Day 169 | 0.93 [0.89 to 0.97] | 0.93 [0.90 to 0.97]

5. Secondary Outcome: Maximum Peak Observed Concentration (Cmax) of LMB763
Description: Pharmacokinetic (PK) parameters were calculated based on LMB763 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC-MS/MS) method. Cmax was determined using non-compartmental methods. No methods for imputation of missing data were used.
Time Frame: pre-dose and 1, 2, 4 and 6 hours after LMB763 administration on Day 1 and Day 14
Population: Pharmacokinetics (PK) analysis set
Measure: Mean (Standard Deviation); unit: Nanogram/milliliter
Arm/Group | LMB763
Number analyzed (Participants) | 41
Nanogram/milliliter
  Day 1 | 1090 (665)
  Day 14: number analyzed (Participants) | 37
  Day 14 | 1300 (691)

6. Secondary Outcome: Time to Reach Maximum Blood Concentrations (Tmax) of LMB763
Description: Pharmacokinetic (PK) parameters were calculated based on LMB763 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC-MS/MS) method. Tmax was determined using non-compartmental methods. Actual time of sample collection was used (not the nominal time point as per scheduled assessment). No methods for imputation of missing data were used.
Time Frame: pre-dose and 1, 2, 4 and 6 hours after LMB763 administration on Day 1 and Day 14
Population: Pharmacokinetics (PK) analysis set
Measure: Median (Full Range); unit: Hour
Arm/Group | LMB763
Number analyzed (Participants) | 41
Hour
  Day 1 | 3.25 [0.75 to 6]
  Day 14: number analyzed (Participants) | 37
  Day 14 | 2 [0 to 6]

7. Secondary Outcome: Area Under the Blood Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast) of LMB763
Description: Pharmacokinetic (PK) parameters were calculated based on LMB763 blood concentrations determined by a validated liquid chromatography and tandem mass spectrometry (LC-MS/MS) method. AUClast was determined using non-compartmental methods. No methods for imputation of missing data were used.
Time Frame: pre-dose and 1, 2, 4 and 6 hours after LMB763 administration on Day 1 and Day 14
Population: Pharmacokinetics (PK) analysis set
Measure: Mean (Standard Deviation); unit: Hour*nanogram/milliliter
Arm/Group | LMB763
Number analyzed (Participants) | 41
Hour*nanogram/milliliter
  Day 1 | 3710 (2510)
  Day 14 | 4850 (2910)

8. Secondary Outcome: Ratio to Baseline in Free Water Clearance
Description: The free water clearance (mL/min) was calculated using the following formula: (Total Volume (mL) / Elapsed Date & Time (min)) * (1-24 hr Urine Osmolality (mOsmol/kg)/ Serum Osmolality (mOsmol/kg))
  The result of free water clearance was rounded to one decimal place prior to statistical analysis. An analysis of covariance (ANCOVA) with treatment as the classification factor and log-transformed baseline as the covariate was conducted for log-transformed ratio to baseline free water clearance. Baseline is the last measurement prior to treatment administration. No methods for imputation of missing data were used. Values reported were back-transformed to original scale. A higher score in the ratio to baseline indicates improvement.
Time Frame: Baseline and day 169
Population: Pharmacodynamics (PD) analysis set. Only participants with a value at both baseline and at Day 169 were included.
Measure: Least Squares Mean (80% Confidence Interval); unit: Ratio
Arm/Group | LMB763 | Placebo
Number analyzed (Participants) | 8 | 11
Ratio | 0.97 [0.86 to 1.10] | 0.97 [0.88 to 1.08]

9. Secondary Outcome: Ratio to Baseline in Lipoprotein A at Day 85
Description: Lipoprotein A (gram/liter) is a component of the lipid profile which is a panel of blood tests used to find abnormalities in lipids. Ratio to baseline in Lipoprotein A was analyzed on a log-scale fitting a repeated measures mixed model including treatment and visit as fixed effects and log of baseline as continuous covariate. Baseline is the last measurement prior to treatment administration. No methods for imputation of missing data were used. Values reported were back-transformed to original scale. A lower score in the ratio to baseline indicates improvement.
Time Frame: Baseline and day 85
Population: as for outcome 4
Measure: Least Squares Mean (80% Confidence Interval); unit: Ratio
Arm/Group | LMB763 | Placebo
Number analyzed (Participants) | 19 | 24
Ratio | 0.72 [0.67 to 0.77] | 0.95 [0.90 to 1.01]

10. Secondary Outcome: Ratio to Baseline in Lipoprotein A at Day 169
Description: as for outcome 9
Time Frame: Baseline and day 169
Population: as for outcome 4
Measure: Least Squares Mean (80% Confidence Interval); unit: Ratio to baseline
Arm/Group | LMB763 | Placebo
Number analyzed (Participants) | 12 | 19
Ratio to baseline | 0.75 [0.66 to 0.85] | 0.89 [0.81 to 0.99]

11. Secondary Outcome: Percent Change From Baseline in Weight
Description: Change from baseline in weight was analyzed on a log-scale fitting a repeated measures mixed model including treatment and visit as fixed effects and log of baseline as continuous covariate. Baseline is the last measurement prior to treatment administration. No methods for imputation of missing data were used. Values reported were back-transformed to original scale. A negative score in the percent change from baseline indicates improvement.
Time Frame: Baseline and days 14, 29, 57, 85, 113, 141 and 169
Population: as for outcome 4
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent change
Arm/Group | LMB763 | Placebo
Number analyzed (Participants) | 41 | 41
Percent change
  Day 14: number analyzed (Participants) | 39 | 41
  Day 14 | -0.08 [-0.45 to 0.29] | -0.13 [-0.50 to 0.23]
  Day 29: number analyzed (Participants) | 37 | 38
  Day 29 | -0.57 [-0.99 to -0.14] | -0.03 [-0.45 to 0.39]
  Day 57: number analyzed (Participants) | 34 | 34
  Day 57 | -0.69 [-1.35 to -0.04] | -0.24 [-0.90 to 0.41]
  Day 85: number analyzed (Participants) | 29 | 34
  Day 85 | -0.41 [-1.21 to 0.38] | 0.08 [-0.70 to 0.86]
  Day 113: number analyzed (Participants) | 25 | 29
  Day 113 | -0.51 [-1.42 to 0.40] | 0.21 [-0.67 to 1.09]
  Day 141: number analyzed (Participants) | 23 | 26
  Day 141 | -0.80 [-1.69 to 0.09] | 0.43 [-0.44 to 1.29]
  Day 169: number analyzed (Participants) | 22 | 28
  Day 169 | -0.61 [-1.60 to 0.39] | 0.55 [-0.38 to 1.47]

12. Secondary Outcome: Percent Change From Baseline in Body Mass Index (BMI)
Description: BMI was determined by height and weight measurements: Body weight (kg)/ [Height (m)]^2. Change from baseline in BMI was analyzed on a log-scale fitting a repeated measures mixed model including treatment and visit as fixed effects and log of baseline as continuous covariate. Baseline is the last measurement prior to treatment administration. No methods for imputation of missing data were used. Values reported were back-transformed to original scale. A negative score in the percent change from baseline indicates improvement.
Time Frame: Baseline and days 14, 29, 57, 85, 113, 141 and 169
Population: as for outcome 4
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent change
Arm/Group | LMB763 | Placebo
Number analyzed (Participants) | 41 | 41
Percent change
  Day 14: number analyzed (Participants) | 39 | 41
  Day 14 | -0.01 [-0.12 to 0.10] | -0.05 [-0.16 to 0.06]
  Day 29: number analyzed (Participants) | 37 | 38
  Day 29 | -0.19 [-0.32 to -0.05] | -0.02 [-0.15 to 0.12]
  Day 57: number analyzed (Participants) | 34 | 34
  Day 57 | -0.23 [-0.44 to -0.02] | -0.07 [-0.28 to 0.14]
  Day 85: number analyzed (Participants) | 29 | 34
  Day 85 | -0.13 [-0.40 to 0.13] | 0.03 [-0.22 to 0.29]
  Day 113: number analyzed (Participants) | 25 | 29
  Day 113 | -0.18 [-0.47 to 0.12] | 0.07 [-0.21 to 0.35]
  Day 141: number analyzed (Participants) | 23 | 26
  Day 141 | -0.31 [-0.60 to -0.01] | 0.16 [-0.12 to 0.45]
  Day 169: number analyzed (Participants) | 22 | 28
  Day 169 | -0.29 [-0.61 to 0.04] | 0.16 [-0.15 to 0.47]

13. Secondary Outcome: Change From Baseline in Waist-to-hip Ratio
Description: Waist-to-hip ratio was derived using waist circumference and hip circumference, which was measured at the greatest protrusion of the buttocks. Change from baseline in waist-to-hip ratio was analyzed on a log-scale fitting a repeated measures mixed model including treatment and visit as fixed effects and log of baseline as continuous covariate. Baseline is the last measurement prior to treatment administration. No methods for imputation of missing data were used. Values reported were back-transformed to original scale. A negative score in the change from baseline indicates improvement.
Time Frame: Baseline and days 14, 29, 57, 85, 113, 141 and 169
Population: as for outcome 4
Measure: Least Squares Mean (80% Confidence Interval); unit: Ratio
Arm/Group | LMB763 | Placebo
Number analyzed (Participants) | 41 | 41
Ratio
  Day 14: number analyzed (Participants) | 39 | 41
  Day 14 | -0.00 [-0.01 to 0.00] | -0.00 [-0.01 to 0.00]
  Day 29: number analyzed (Participants) | 37 | 37
  Day 29 | -0.00 [-0.01 to 0.00] | 0.00 [-0.00 to 0.01]
  Day 57: number analyzed (Participants) | 34 | 34
  Day 57 | -0.00 [-0.01 to 0.00] | 0.00 [-0.01 to 0.01]
  Day 85: number analyzed (Participants) | 29 | 34
  Day 85 | -0.00 [-0.01 to 0.00] | 0.01 [-0.00 to 0.01]
  Day 113: number analyzed (Participants) | 25 | 29
  Day 113 | -0.00 [-0.01 to 0.01] | 0.01 [0.00 to 0.02]
  Day 141: number analyzed (Participants) | 24 | 26
  Day 141 | -0.00 [-0.01 to 0.01] | 0.02 [0.01 to 0.03]
  Day 169: number analyzed (Participants) | 22 | 28
  Day 169 | -0.00 [-0.01 to 0.01] | -0.00 [-0.01 to 0.00]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the start of treatment to 28 days after end of treatment, assessed up to maximum duration of 197 days
Description: Any sign or symptom that occurs during the study treatment plus the 28 days post treatment
Groups:
- Total: Total
Arm/Group | LMB763 | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/42 | 0/83
Serious Adverse Events (participants affected / at risk) | 2/41 | 2/42 | 4/83
Other Adverse Events (participants affected / at risk) | 28/41 | 23/42 | 51/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LMB763 (N=41) | Placebo (N=42) | Total (N=83)
Erysipelas (Infections and infestations) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Renal disorder (Renal and urinary disorders) | 0 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LMB763 (N=41) | Placebo (N=42) | Total (N=83)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 3
Colitis (Gastrointestinal disorders) | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 1 | 1 | 2
Fatigue (General disorders) | 2 | 0 | 2
Oedema peripheral (General disorders) | 1 | 0 | 1
Pain (General disorders) | 1 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 1
Acarodermatitis (Infections and infestations) | 1 | 1 | 2
Adenoviral conjunctivitis (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 2 | 2
Erysipelas (Infections and infestations) | 1 | 1 | 2
Gastroenteritis (Infections and infestations) | 2 | 1 | 3
Influenza (Infections and infestations) | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 2 | 3
Sinusitis (Infections and infestations) | 1 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 3
Urinary tract infection bacterial (Infections and infestations) | 1 | 1 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Blood bicarbonate decreased (Investigations) | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 4 | 3 | 7
Blood fibrinogen increased (Investigations) | 0 | 1 | 1
Blood glucose increased (Investigations) | 1 | 0 | 1
Blood pressure increased (Investigations) | 0 | 2 | 2
Blood uric acid increased (Investigations) | 1 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 1 | 1
Serum ferritin decreased (Investigations) | 0 | 1 | 1
Ultrasound scan abnormal (Investigations) | 1 | 0 | 1
Urine albumin/creatinine ratio increased (Investigations) | 0 | 3 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cerebral artery stenosis (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 2 | 2 | 4
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1
Sciatica (Nervous system disorders) | 1 | 1 | 2
Somnolence (Nervous system disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 1
Pruritus genital (Reproductive system and breast disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 6 | 19
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 2 | 4
Hypotension (Vascular disorders) | 1 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT03804879/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT03804879/SAP_001.pdf